CLINICAL TRIAL: NCT05697679
Title: Effects of a Physical Activity Promotion Program on Body Composition in Emerging Adults With Physical Inactivity: A Study Protocol of a Randomized Controlled Trial
Brief Title: Effects of Physical Activiy Promotion Intervention Programs in Emerging Adulthood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Tao (Other)
Responsible Party: Sponsor-Investigator, Xu Tao, Principal Investigator, Hangzhou Normal University
Organization: Hangzhou Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022059
Record Dates: First submitted 2022-12-29; First posted 2023-01-26 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Body Composition; Health Behavior
Keywords: Body composition; Theory of goal attainment; Eating behavior; Health behavior
MeSH Terms: conditions — Health Behavior; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The present study is based on a stratified randomized controlled design with two groups. The stratification is done with four groups based on the BMI (underweight, ≤18.5; normal weight, 18.5-24.0; overweight, 24.0-28.0; obesity, BMI of 28 or greater) indicated at registration. Each participant is randomly assigned to either the different group 1 week before the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The first author will use randomizer.org for randomization. Recruitment without informing the subjects of study participation and group allocation to blind the subjects. And the allocation is also concealed for researchers in charge of data collection and processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual management group (Experimental): The intervention group is intervened with the TG
  Interventions: Behavioral: Treatment group
- Goal-attainment-theory-based self-management group (Active Comparator): The group is intervened with the CG
  Interventions: Behavioral: Contral group

INTERVENTIONS:
Behavioral: Treatment group — WeChat groups will be set up, and once a week on Monday, articles on physical exercise and once a week on Wednesday, 3-minute films about health education will be shared. For the duration of the 3-month intervention period, the following technologies will be used to deliver the GAT-pap: (1) Short Messaging Service (SMS) text (batch messaging); (2) WeChat (e.g., physical activity guidelines, group chats); and (3) monthly face-to-face interviews (behaviour change promotion, risk factor management). Although not essential, participants will be urged to register their daily exercise in the group chat. In order to determine if they are accomplishing their goals and what objectives they should be pursuing, the researchers will develop customised training regimens for each participant.
  Other Names: TG
  Arms: Usual management group
Behavioral: Contral group — One or two times each week, participants in the control group will get general lifestyle advice through SMS. They will not participate in the intervention's fitness routines, online classes, group chats, or films with health educators. Individual workout regimens, goals, or comments are not given by researchers. Participants in the control group's complaints or questions will always be answered with basic health information and suggestions. Researchers won't ask for individual advice or comments from other professionals.
  Other Names: CG
  Arms: Goal-attainment-theory-based self-management group

SUMMARY:
This is a prospective, double-blinded, 16-week, randomized controlled trial (RCT). Young adults aged 18-25 years are recruited in this study. Based on King's (1981) goal attainment theory, a diet-exercise program is created. The aim of this study is to investigate the impact of physiological indicators and health behaviours by conducting an exerciset programme and intensive therapy.

DETAILED DESCRIPTION:
Background:

Emerging adulthood (18-25 years), has been linked to increased probability of unhealthy and risky lifestyle behaviours, such as alcohol, tobacco and other drug use, dangerous driving, unprotected sex, and unhealthy dietary choices. These lifestyle behaviours are associated with some of the key leading causes of premature death and disease burden in this age group. Thus, reducing the prevalence of risky and unhealthy lifestyle behaviours among emerging adults is a priority for health promoters and governments.

Aim:

The researchers hypothesize that a health program based on King's goal achievement theory have a significant effect on body composition among college students. Therefore, in this study, researchers will explore the impact of a health program based on King's goal achievement theory on the body composition of college students.

Methods:

This is a prospective, double-blinded, 12-week, randomized controlled trial in Hangzhou. Participants are randomly allocated in a 1:1 ratio to two groups using blocked randomization. WeChat groups will be set up, and once a week on Monday, articles on physical exercise and once a week on Wednesday, 3-minute films about health education will be shared. For the duration of the 3-month intervention period, the following technologies will be used to deliver the GAT-pap: (1) Short Messaging Service (SMS) text (batch messaging); (2) WeChat (e.g., physical activity guidelines, group chats); and (3) monthly face-to-face interviews (behaviour change promotion, risk factor management). Although not essential, participants will be urged to register their daily exercise in the group chat. In order to determine if they are accomplishing their goals and what objectives they should be pursuing, the researchers will develop customised training regimens for each participant.

Participants and demographic data:

Healthy individuals with a sedentary lifestyle will be recruited to participate in the study through online and print advertisements posted at Hangzhou Normal University (Hangzhou, China) and surrounding communities. Sedentary behavior is defined as any waking behavior characterized by an energy expenditure ≤ 1.5 metabolic equivalents, such as sitting, reclining or lying down. The participants are able to express themselves and to individually complete the International Physical Activity Questionnaire (IPAQ)

Procedure and Data collection:

This is a prospective, double-blinded, 16-week, randomized controlled trial (RCT) complied with the ethical principles of the Helsinki Declaration and the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) checklist. It was approved by the Medical Ethical Committee of the Hangzhou Normal University (Ratification date is November 14, 2022, 2022059)

Statistical analysis:

This study will employ Predictive Analytics Suite Workstation (IBM SPSS 28.0) to analyze the collected data. The data analyses will include demographic variables and the scores of IPAQ, SBES at the interval of 12 weeks of all of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Having a sedentary lifestyle. ( Sedentary behavior is defined as any waking behavior characterized by an energy expenditure ≤ 1.5 metabolic equivalents, such as sitting, reclining or lying down. )

Exclusion Criteria:

* Diabetes
* Cardiovascular disease risk
* Upper respiratory infection
* Smoking
* Injury or disease that limited exercise ability
* Using of any medication within the last 3 months
* Lactose intolerance
* Celiac diseas
* Food allergies
* Specific dietary regiments (e.g., vegetarian diet, intermittent fasting or less common diets)
* Pregnancy or planning pregnancy during the study period.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in body composition | Before and 16 weeks after the intervention
  Participants will have body composition measured by using bioelectrical impedance analysis (BIA) with InBody 720 device. According to the InBody device manufacturer's testing procedures, participants will be told not to exercise for at least 24 hours before the test, not to consume alcohol or excessive amounts of caffeine, and not to eat and drink for four hours before the test, but water can be consumed up to 45 minutes before the test.

SECONDARY OUTCOMES:
Changes in amount of physical activety | Before and 16 weeks after the intervention
  The International Physical Activity Questionnaire-Short Form (IPAQ-SF) prepared by the International Working Group on Physical Activity Measurement, was selected to investigate the physical activity levels. The IPAQ has been translated into Chinese with a good reliability and validity. There are 7 items in the questionnaire. Three intensities of physical activities during the last seven days were collected, including (1) vigorous-intensity activities such as speed swimming or playing basketball, (2) moderate-intensity activities such as slow dancing or strenuous household chores, and (3) low-intensity activities such as walking. Each activity had its own metabolic equivalent (MET) energy expenditure, and the vigorous-, moderate-, and low-intensity activities equaled 8.0, 4.0, and 3.3 METs. The amount of physical activity was estimated by weighting the intensity and time spent performing each activity with its MET.
Changes in self-efficacy | Before and 16 weeks after the intervention
  The Simplified Chinese version of the Health-Related Diet and Exercise Self-Efficacy Scale (HRDESES) included 8 items under 2 dimensions: diet subscale and exercise subscale. Response options are rated on a 5-point scale: 0 (I'm not sure), 1 (mostly I cannot), 2 (don't know), 3 (mostly I can), or 4 (I'm sure I can). The total score ranges from 0 to 32, with a higher score indicating higher levels of health-related diet and exercise self-efficacy. The Cronbach's α of the HRDESES was 0.87 for the total scale, 0.86 for the diet The simplified Chinese version of the health-related diet and exercise self-efficacy scale subscale and 0.91 for the exercise subscale
Motivation level | Before and 16 weeks after the intervention
  Measurement of changes in motivation levels will be applied using the Treatment Self-Regulation Questionnaire (TSRQ) created by Ryan

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xu, Principal Investigator — Hangzhou normal univesity
Locations (1):
- Hangzhou Normal University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu T, Liu CY, Tao YX, Cai XT, Wu YY, Chen R, Xiao T, Liu MY. Effects of a goal attainment theory-based intervention on physical activity, body composition, and motivation in emerging adults with physical inactivity: A randomized controlled trial. Public Health. 2025 Jan;238:280-288. doi: 10.1016/j.puhe.2024.12.007. Epub 2024 Dec 19. PMID 39706105
- [Derived] Xu T, Tao Y, Chen R, Strachan G, Cai X, Liu C. Effects of a physical activity promotion programme on body composition in emerging adults with physical inactivity: a study protocol of a randomised controlled trial. BMJ Open. 2023 Oct 5;13(10):e076123. doi: 10.1136/bmjopen-2023-076123. PMID 37798029